CLINICAL TRIAL: NCT06048562
Title: Incidence of Hypertrophic Cardiomyopathy in Infants of Diabetic Mothers Attending in NICU
Brief Title: Incidence of Hypertrophic Cardiomyopathy in Infants of Diabetic Mothers Attending in NICU at Assiut University Children Hospital During One Year
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelkareem, Assuit university, Assiut University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: hypertrophic cardiomyopathy
Record Dates: First submitted 2023-09-16; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Echocardiography

STUDY DESIGN:
Intervention Model Description: To evaluate all full term infants of diabetic mother for the presence of hypertrophic cardiomyopathy who admitted in NICU at Assiut University Children Hospital and to follow up of these cases after 6 months for recovery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- idm (Experimental): evaluation idm for cardiomyopathy
  Interventions: Diagnostic Test: echocardiography

INTERVENTIONS:
Diagnostic Test: echocardiography — evaluation idm for cardiomyopathy by echo

SUMMARY:
To evaluate all full term infants of diabetic mother for the presence of hypertrophic cardiomyopathy who admitted in NICU at Assiut University Children Hospital and to follow up of these cases after 6 months for recovery.

DETAILED DESCRIPTION:
Diabetes is the most common endocrine disorder complicating pregnancy. Incidence of both type-I and type-II diabetes is increasing, throughout the world. As the incidence of diabetes continues to rise and increasingly affects individuals of all ages including young adults and children, women in child bearing age are at increased risk of diabetes during pregnancy [1].

The type 1 diabetes around the time of conception produces marked risk of embryopathy (neural tube defects, cardiac defects, and caudal regression syndrome) as these mother have high glycosylated hemoglobin at the time of embryogenesis (around 6-8 weeks of gestation) rather than IDM that are born to type 2 diabetes mothers who have macrosomia and other milder problems. The mothers who have been diagnosed as severe and unstable type1 diabetes in the later part of gestation have high chances of neonate being more affected with intrauterine growth restriction, asphyxia, and fetal death [2] and [3].

Due to the teratogenic effect of maternal diabetes, the reported incidence of congenital malformations among the newborns of diabetic mothers is five times greater than that of the general population [4].

Cardiac malformations are one of the most common types of these malformations which occur in about 8.5% of cases that is about 10 times more than its incidence in normal population (0.8%) [5].

Fetuses exposed to maternal hyperglycemia and hyperinsulinism, are prone to develop hypertrophic cardiomyopathy. It primarily affects the inter-ventricular septum, but can extend to the myocardium in more severe cases. Although the perinatal mortality rates associated with diabetes in pregnancy have declined considerably during the past eight decades and are now near those in the general population, it is only through continuing vigilance that such advances can be maintained. Both fetal and neonatal deaths occurred with increased frequency in diabetic pregnancies before the advent of modern management methods, and fetal deaths nationwide continue to be significantly higher among diabetic than non-diabetic pregnancies [6].

The most recent available data indicate that the relative risk of stillbirth in pregnancies complicated by type 1 diabetes (compared to the general population) is 2.9-4.3 folds, and for type 2 diabetes 2.5-4.5 fold [7].

ELIGIBILITY:
Inclusion Criteria:

* all infants of diabetic mothers were admitted at NICU

Exclusion Criteria:

* NO

Ages: 6 Hours to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
evaluate hypertrophic cardiomyopathty in IDM | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abdelkareem, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang J, Cummings EA, O'connell C, Jangaard K. Fetal and neonatal outcomes of diabetic pregnancies. Obstet Gynecol. 2006 Sep;108(3 Pt 1):644-50. doi: 10.1097/01.AOG.0000231688.08263.47. PMID 16946226
- [Background] [3] Correa A, Gilboa SM, Besser LM, Botto LD, Moore CA, Hobbs CA, etal, Diabetes mellitus and birth defects. Obstetric Anesthesia Digest. 2009 Mar 1;29(1):40-1.
- [Result] Hunt KJ, Schuller KL. The increasing prevalence of diabetes in pregnancy. Obstet Gynecol Clin North Am. 2007 Jun;34(2):173-99, vii. doi: 10.1016/j.ogc.2007.03.002. PMID 17572266